CLINICAL TRIAL: NCT06732895
Title: A Phase 2b, Multicenter, Double-Blind, Randomized, Placebo-controlled Trial Evaluating Efficacy and Safety of Subcutaneous Doses of Navepegritide Administered Once Weekly for 52 Weeks in Adolescents (12-18 Years of Age) With Achondroplasia.
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of Navepegritide in Adolescents (12 - 18 Years of Age) With Achondroplasia.
Acronym: teACH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASND0045; 2024-514208-15-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Navepegritide (Experimental): Once weekly double-blinded treatment with SC injection of 100 µg/kg of navepegritide for 52 weeks
  Interventions: Drug: Navepegritide
- Placebo for Navepegritide (Placebo Comparator): Once weekly double-blinded treatment with SC injection of 100 µg/kg of placebo for navepegritide for 52 weeks
  Interventions: Drug: Placebo for navepegritide

INTERVENTIONS:
Drug: Navepegritide — Once-weekly subcutaneous injection of 100 µg/kg navepegritide for 52 weeks
  Arms: Navepegritide
Drug: Placebo for navepegritide — Once-weekly subcutaneous injection of 100 µg/kg placebo for navepegritide
  Arms: Placebo for Navepegritide

SUMMARY:
The purpose of this clinical trial is to evaluate efficacy and safety of once weekly subcutaneous (SC) doses of navepegritide 100 μg/kg compared to placebo (inactive drug) in adolescents aged 12 to 18 years with Achondroplasia. What will be measured is Annualized Growth Velocity after a 52-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent and/or assent of the participant, participant parent(s) or legal guardian(s) of the participant, and as required by the institutional review board/human research ethics committee/independent ethics committee (IRB/HREC/IEC). For participants who are below the age of consent, a written assent will be obtained in accordance with applicable requirements as required by IRB/HREC/IEC. Upon reaching the legal age of consent, depending on applicable requirements, these participants will be asked to give their own written consent.
* Male or female, between 12 (inclusive) and 18 years of age at the time of randomization
* Clinical diagnosis of ACH with documented genetic confirmation available. Documentation of historic test results are acceptable for proof of diagnosis.
* Parent(s)/legal guardian(s) willing and able to administer weekly SC injections of IMP and to follow the protocol.
* At least one historical standing height measurement available from medical records. The measurement must have been collected between 6 months to 15 months prior to the time of screening.

Exclusion Criteria:

* Participation (signed informed consent) in any interventional clinical trial within 3 months prior to Screening unless no doses of IMP was given.
* Decreased growth velocity (AGV less than 1.5 cm/year based on measurement over a period of at least 6 months) or radiological evidence of growth plate closure.
* Known or suspected hypersensitivity to the IMP or related products (trehalose, tris[hydroxymethyl]aminomethane, succinate, and mPEG).
* Have a growth disorder or medical condition other than ACH that results in short stature, or abnormal growth such as SADDAN, hypochondroplasia, growth hormone deficiency, Turner syndrome, pseudo-ACH, inflammatory bowel disease, celiac disease, hypothyroidism, hyperthyroidism, or diabetes mellitus.
* Severe mutation in the FGFR3 gene, e.g. two variants on the same allele or severe ACH with developmental delay and acanthosis nigricans, are not eligible for trial participation.
* Have received any dose of prescription medications and/or IMP (placebo treatment only is allowed, if documented) or surgical intervention intended to affect stature, growth, or body proportionality at any time.
* Requires, or anticipated to require, chronic (more than 4 weeks) or repeated treatment (more than twice/year and less than 3 weeks/year) with systemic corticosteroids during participation in the trial. Chronic use of high dose inhaled corticosteroids is not allowed.
* Known history of presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones.
* Known history of any bone-related surgery affecting growth potential of long bones, such as:

  * Orthopedic reconstructive surgery for bone lengthening (e.g., procedures for leg bowing such as 8-plate are not exclusionary).
  * Ventriculoperitoneal (VP) shunt and laminectomy with full recovery are allowed with minimum of 6 months of bone healing.
  * Bone fracture within 6 months prior to screening (within 2 months for fracture of digits and buckle fractures).
* Clinically significant findings at Screening, such as:

  * Expected to require surgical intervention during participation in the trial that may significantly affect trial parameters (confounding of safety events) or would prevent the participant from performing trial procedures. Common surgeries, such as insertion of grommets, adenoidectomy, tonsillectomy, or myringotomy tube placement, are permitted.
  * Severe untreated sleep apnea or newly initiated sleep apnea treatment (e.g., Continuous Positive Airway Pressure [CPAP] in the previous 2 months prior to Screening.
  * MS disease, such as Salter-Harris fractures or clinical and/or radiographic evidence of severe hip pathology
  * Otherwise, are considered by the Investigator to be unfit to receive trial treatment or undergo trial related procedures.
* Have a clinically significant finding or arrhythmia as determined by the investigator in consultation with the medical monitor that indicates abnormal cardiac function or conduction that includes, but is not exclusive to:

  * Repaired or unrepaired coarctation.
  * Moderate or greater complexity congenital heart disease including tetralogy of Fallot, Atrioventricular septal defects, truncus arteriosus, total anomalous pulmonary venous return, double outlet right ventricle, or single ventricle heart disease.
* QT corrected using Fridericia's correction (QTcF) ≥ 450 msec at Screening.
* Known history or presence of condition that impacts hemodynamic stability (such as autonomic dysfunction and orthostatic intolerance).
* Known history or presence of the following:

  * Chronic anemia (iron deficiency anemia that is resolved or adequately treated in the Investigator's opinion is allowed).
  * Chronic renal insufficiency defined as estimated glomerular filtration rate (eGFR) according to the revised bedside Schwartz equation less than 60 mL/min/1.73 m2 for more than 3 months.
  * Chronic or recurrent illness that can affect hydration or volume status, including conditions associated with decreased nutritional intake or increased volume loss.
* Known history or presence of malignant disease.
* Participant with serum 25-hydroxy-vitamin D (25OHD) levels of less than 30 nmol/L (less than 12 ng/mL) at Screening Visit will be excluded. Participants with 25OHD levels between 30-50 nmol/L (12-20 ng/mL) can be randomized provided treatment with Vitamin D supplementation is initiated according to local standards.
* Any disease or condition that, in the opinion of the Investigator, may make the participant unlikely to fully complete the trial, may confound interpretation of trial results, or may present undue risk from receiving trial treatment. This could include family situations, complications or manifestations, or medications that might impact safety or be considered confounding.
* Sexually active male and female participants and female partners of male participants of childbearing potential not using a highly effective form of contraceptive for the entire trial period and for 90 days after last dose of trial treatment.
* Female participants who are pregnant, lactating or breastfeeding.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Growth Velocity | 52 weeks
  cm per year

SECONDARY OUTCOMES:
Height Z-score | 52 weeks
  Number of standard deviations

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Ascendis Pharma A/S
Locations (5):
- Ascendis Investigational Site, Montreal, Canada
- Ascendis Investigational Site, Copenhagen, Denmark
- Ascendis Investigational Site, Paris, France
- Ascendis Investigational Site, Dublin, Ireland
- Ascendis Investigational Site, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No